CLINICAL TRIAL: NCT04377737
Title: Incidence of Covid-19 in School Children During the Pandemic Period in Nice
Brief Title: Incidence of Covid-19 in School Children
Acronym: COVIDECOLE
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Human Subjects Protection Review: submitted, denied
Sponsor: Fondation Lenval (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 20-HPNCL-02
Record Dates: First submitted 2020-05-04; First posted 2020-05-06 (Actual); Last update posted 2020-05-27 (Actual); Status verified 2020-05

CONDITIONS: Infection; Viral, Coronavirus
Keywords: Covid19; Incidence; School; Pandemia; Children
MeSH Terms: conditions — Coronavirus Infections; COVID-19 | interventions — COVID-19 Nucleic Acid Testing

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RT-PCR Covid-19 (Other)
  Interventions: Diagnostic Test: RT-PCR Covid-19

INTERVENTIONS:
Diagnostic Test: RT-PCR Covid-19 — estimation of the prevalence of positive rt-PCR in school children during the pandemic period

SUMMARY:
The Coronavirus disease 2019 (COVID-19) is causing a global pandemic with high morbidity and mortality among adults and mainly the elderly. Children seem to be little or not affected by this infection. It is estimated that children could be asymptomatic or pauci-symptomatic carriers and thus be vectors of the disease. This is why measures to close schools and confine populations have been decreed in a large number of countries, including France. However, there are only a few data on the prevalence of COVID19 disease in children. The deconfinement strategy depends on data on the prevalence of the disease, especially in children.

Investigators propose to evaluate the incidence of Covid-19 in preschool and elementary schools children in the city of Nice (South of France) during the pandemic period using a local prospective study of 914 children

DETAILED DESCRIPTION:
The Coronavirus disease 2019 (COVID-19) is causing a global pandemic with high morbidity and mortality among adults and mainly the elderly. Children seem to be little or not affected by this infection. It is estimated that children could be asymptomatic or pauci-symptomatic carriers and thus be vectors of the disease. However, the role of the children in the spread of COVID-19 injection remains unclear.

Measures to close schools and to confine populations have been decreed in a large number of countries, including France. This decision has been based on epidemiologic data of other viral infections having droplet transmission and on data of Middle East Respiratory Syndrome-related coronavirus (MERS-CoV) asymptomatic portage.

Furthermore, there are only a few data on the prevalence of COVID19 disease in children. The deconfinement strategy depends on data on the prevalence of the disease, especially in children.

Therefore, investigators propose to evaluate the incidence of Covid-19 in preschool and elementary schools children in the city of Nice (South of France) during the pandemic period using a local prospective study of 914 children.

This study will start on 11th May 2020, date of school reopening, in order to collect epidemiologic data about Covid-19 carriage among schoolers and to support governmental strategy for the new school year in September 2020.

ELIGIBILITY:
Inclusion Criteria:

Age ranging from 3 to 10 years old

* Children attending to school in Nice
* Informed consent
* French insurance subscribed

Exclusion Criteria:

* Refusal to participate from the parents or the child
* Bleeding disorders

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2020-05-15 (Estimated); Primary Completion 2020-08 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
evaluation of the prevalence of positive real-time-polymerase chain reaction (rt-PCR) in school children during the pandemic period in Nice | at 42 days
  measure by two rt-PCR COVID-19 tests regardless the serological status of the child

SECONDARY OUTCOMES:
evaluation of the serological prevalence of the Covid-19 infection | at inclusion and at 42 days
  measure by two serological COVID-19 test (IgG and/or IgM)
evaluation of the COVID-19 reinfection among seropositive children at the inclusion time | at inclusion and at 42 days
  measure by two serological COVID-19 test (IgG and/or IgM)
evaluation of the prevalence of positive rt-PCR of other respiratory viruses (including others coronavirus) | at 42 days
  positivity of rt-PCR test for other viruses (adenovirus, metapneumovirus, picornavirus, respiratory syncytial virus, influenza et parainfluenza and other coronavirus strains)
comparison of inflammatory response level between different coronavirus strains | at 42 days
  measure of level of the two inflammation biomarkers (IFIT1 interferon and CCL8)
Estimation of medico-social risk factors associated with COVID-19 infection | at 42 days
  measure of the medico-social relative risk associated with rt-PCR COVID-19 test positivity among : school level, gender, school type, day care facilities before 11th May, number of siblings, housing type, number of bedrooms, precariousness level, by score EPICES ( (Evaluation de la Précarité et des Inégalités de santé dans les Centres d'examens de santé, means Assessment of precariousness and health inequalities in health examination centers).
  Questionnaire of EPICES counts 11 items, the answer to each question is assigned a coefficient, the sum of the 11 answers gives the score EPICES. The score is continuous, it varies from 0 (lack of precariousness) to 100 (maximum precariousness).

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpitaux Pédiatrique de Nice CHU Lenval, Nice, France